CLINICAL TRIAL: NCT02808949
Title: Phase 1 Pharmacokinetic Study of the Dapivirine Vaginal Ring in Lactating Women
Brief Title: Pharmacokinetic Study of the Dapivirine Vaginal Ring in Lactating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTN-029/IPM 039; NCT02658227 (obsolete NCT alias)
Record Dates: First submitted 2015-12-18; First posted 2016-06-22 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: Prevention; Lactating Women; Healthy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Dapivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Age Groups (Experimental): Dapivirine levels in breast milk will be measured in 16 participants. All participants will wear the Dapivirine Vaginal Ring for 14 consecutive days.
  Interventions: Drug: Dapivirine

INTERVENTIONS:
Drug: Dapivirine — Participants will receive a silicone elastomer vaginal matrix ring containing 25 mg of dapivirine to wear for approximately 14 continuous days. Participants age 18 and over, at least 6 weeks postpartum, able to produce and express breast milk for 14 consecutive days.
  Other Names: Dapivirine vaginal ring

SUMMARY:
Phase 1 PK Study of the Dapivirine Vaginal Ring in Lactating Women.

DETAILED DESCRIPTION:
PK Study of the Dapivirine Vaginal Ring in Lactating Women.

ELIGIBILITY:
Inclusion Criteria:

Women must meet all of the following criteria (by self-report, unless otherwise indicated) to be eligible for inclusion in the study:

1. Age 18 or older at screening as verified per site SOP
2. Per participant report, at least 6 weeks postpartum at Enrollment
3. Willing and able to provide written informed consent to be screened for and take part in the study
4. Willing and able to provide adequate locator information, as defined in site SOP
5. Willing and able to communicate in spoken and written English
6. HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in Appendix II and willing to receive HIV test results Note: HIV-1/2 screening may be omitted at Enrollment if the time between Screening and Enrollment is < 30 days
7. Prior to Enrollment, breastfeeding of child has stopped
8. Participant has no intention of providing expressed breast milk to her child(ren) or to others for consumption after initiation of study product Note: Providing stored breast milk to child(ren) that has been expressed prior to study product exposure is not exclusionary
9. Willing and able to express breast milk at least twice daily for the duration of study drug exposure
10. Per participant report, using an effective method of contraception at Enrollment, and intending to continue the use of an effective method for the duration of study participation. Effective methods for MTN-029/IPM 039 include: hormonal methods (except contraceptive VRs), intrauterine device (IUD) inserted at least 28 days prior to enrollment, engages in sex exclusively with women, sterilized (self or partner), or sexually abstinent for the past 90 days
11. Women over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies (Addendum 1 to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, November 2007), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
12. At Screening, participant states a willingness to refrain from receptive sexual activity (including penile-vaginal intercourse, anal intercourse, receptive oral intercourse, finger stimulation) and from inserting any non-study objects into the vagina (including tampons, sex toys, female condoms, diaphragms, menstrual cups, cervical caps or any other vaginal barrier method, etc.), for 24 hours prior to each clinic visit.
13. At Screening, participant states a willingness to refrain from the use of vaginal products, including, spermicides, lubricants, contraceptive VRs, douches, vaginal medications, etc., for the duration of study participation
14. Per participant report at Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, vaccines or breast milk sampling for the duration of study participation Note: Participation in observational studies is not exclusionary

Exclusion Criteria:

Women who meet any of the following criteria (by self-report, unless otherwise indicated) will be excluded from the study:

1. Participant report of any of the following:

   * History of adverse reaction to any component of dapivirine VR
   * Participation in investigational drug or device trial within 30 days prior to the Enrollment Visit (Day 0)
   * Use of vaginal medication(s) 5 days prior to Enrollment (Day 0)
   * Complication of lactation requiring treatment, e.g., mastitis
2. At the time of Screening and Enrollment, clinical evidence of milk supply less than 1 ounce per expression
3. As determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
4. Grade 2 or higher AST/ALT at Screening Visit:

   Note: Otherwise eligible participants with an exclusionary AST/ALT may be retested during the screening process.
5. Positive urine pregnancy test at screening or enrollment
6. Diagnosed with urinary tract infection (UTI) at Screening or Enrollment Note: Otherwise eligible participants diagnosed with UTI during screening are offered treatment and may be enrolled after completing treatment and all symptoms have resolved.
7. Diagnosed with an STI or a reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines at Screening or Enrollment
8. On pelvic exam, any of the following findings:

   * Incomplete postpartum involution of the uterus
   * Clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff)
9. Use of oral and/or vaginal preparations of antibiotic or antifungal medications within 5 days of Enrollment
10. At Screening or Enrollment, any social or medical condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 14 Days
  To assess the pharmacokinetics of dapivirine vaginal ring used for 14 consecutive days in lactating women

SECONDARY OUTCOMES:
Safety and Tolerability of dapivirine ring in lactating women | 14 days
  To assess safety and tolerability of dapivirine vaginal ring used for 14 consecutive days in lactating women
Adherence to dapivirine vaginal ring use in lactating women | 14 days
  To assess adherence to dapivirine vaginal ring use in lactating women

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hoesley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Alabama CRS, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noguchi LM, Hoesley C, Kelly C, Scheckter R, Bunge K, Nel A, Marzinke MA, Hendrix CW, Dezzutti CS, Hillier SL, Bogen DL, Piper JM, Beigi RH. Pharmacokinetics of Dapivirine Transfer into Blood Plasma, Breast Milk, and Cervicovaginal Fluid of Lactating Women Using the Dapivirine Vaginal Ring. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e01930-18. doi: 10.1128/AAC.01930-18. Print 2019 Mar. PMID 30602513